CLINICAL TRIAL: NCT05249816
Title: An Observer-Blinded Phase 3 Study to Evaluate the Safety and Immunogenicity of a Single Booster of the NVX-CoV2373 Vaccine in Adults Previously Vaccinated With the BBIBP-CorV Vaccine
Brief Title: Phase 3 Boosting Study for the SARS-CoV-2 rS Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cogna Technology Solutions LLC (Industry)
Collaborators: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: G42-HC-2021001
Record Dates: First submitted 2022-02-18; First posted 2022-02-22 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
MeSH Terms: interventions — NVX-CoV2373 adjuvated lipid nanoparticle; BIBP COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVX-CoV2373 (Experimental): NVX-CoV2373 (5 μg): Coformulated prototype SARS-CoV-2 rS vaccine with Matrix-M adjuvant: supplied as a solution for preparation for injection, at a concentration of 10 μg antigen and 100 μg adjuvant per mL. The vaccination regimen will comprise of 1 intramuscular (IM) injection on Day 0 of 0.5 mL injection volume at a dose of 5 μg of antigen with 50 μg Matrix-M adjuvant.
  Interventions: Biological: NVX-CoV2373
- BBIBP CorV (Active Comparator): Sinopharm BBIBP-CorV vaccine administered per manufacturer instructions as a single intramuscular injection.
  Interventions: Biological: BBIBP-CorV vaccine

INTERVENTIONS:
Biological: NVX-CoV2373 — A single booster injection of NVX-CoV2373 with Matrix-M adjuvant. 0.5 mL injection volume at a dose of 5μg of antigen with 50 μg Matrix-M adjuvant
  Other Names: Novavax
  Arms: NVX-CoV2373
Biological: BBIBP-CorV vaccine — BBIBP-CorV vaccine administered per manufacturer instructions.
  Other Names: Sinopharm BBIBP-CorV
  Arms: BBIBP CorV

SUMMARY:
This is an observer-blinded Phase 3 study to evaluate the safety and immunogenicity of a single booster dose of the Novavax severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) recombinant (r) spike (S) protein nanoparticle vaccine adjuvanted with Matrix-MTM (NVX-CoV2373) in adults previously vaccinated with the BBIBP-CorV vaccine. The study will enroll approximately1,000 participants >18 years of age. All participants will be randomized in a 1:1 ratio to receive a single booster dose of NVX-CoV2373 or the BBIBP-CorV vaccine. All participants will receive the booster dose on Day 0 and remain on study for immunogenicity and safety data collection through Day 180. An interim analysis will be performed of safety and immunogenicity data gathered through Day 28.

DETAILED DESCRIPTION:
Novavax, Inc., is developing recombinant vaccines adjuvanted with the saponin-based Matrix-M for the prevention of disease caused by SARS-CoV-2. Both nonclinical and clinical data to date (Liu 2011; Keech 2020; Formica 2021; Heath 2021) support continued clinical development of SARS-CoV-2 rS vaccines combined with Matrix-M adjuvant as potential vaccines against SARS-CoV-2.

Due to waning immunity following primary vaccination against SARS-CoV-2 as well as the emergence of SARS-CoV-2 variants (eg, Alpha, Beta, Gamma, Delta and Omicron), a number of countries have administered or are planning to administer booster doses of vaccine to either specific subgroups or to their general population. As part of this effort, both homologous boosting (boosting with the same vaccine used for the primary vaccination series) or heterologous boosting (boosting with a vaccine that differs from that used for the primary vaccination series) are being evaluated.

The present study aims to investigate the safety and immunogenicity of a single booster of NVX-CoV2373 administered to participants who have already been immunized with BBIBP-CorV vaccine. The NVX-CoV2373 booster will be administered > 180 days after the second dose of BBIBP-CorV vaccine, and the ability of the vaccine to increase antibody titers against the prototype SARS-CoV-2 strain as well as the ability to induce cross-neutralizing antibodies to variant strains will be evaluated. If favorable immunogenicity and safety profiles are observed following a booster dose of NVX-CoV2373, this option would add flexibility to the global COVID-19 vaccination effort and potentially decrease the need to develop variant-specific vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age, inclusive, at screening.
2. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
3. Females of childbearing potential (defined as any female who has experienced menarche) who is NOT surgically sterile (i.e., hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or postmenopausal (defined as amenorrhea at least 12 consecutive months), must agree to either be heterosexually inactive OR consistently use a medically acceptable method of contraception, from enrollment and to 3 months after the last vaccination. Medically acceptable methods of contraception include:

   1. Condoms (male or female)
   2. Diaphragm with spermicide
   3. Cervical cap with spermicide
   4. Intrauterine device
   5. Oral or patch contraceptives
   6. Norplant®, Depo-Provera®, or other in country regulatory approved contraceptive method that is designed to protect against pregnancy
   7. Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle

      * NOTE: Periodic abstinence (e.g., calendar, ovulation, symptom-thermal, post- ovulation methods) and withdrawal are not acceptable methods of contraception.
      * Condoms (male or female) are not required if a female partner is using an alternative medically acceptable method of contraception as listed in points 3a-g).
4. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges as determined by the investigator prior to the first vaccination.
5. Agrees to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study. NOTE: For participants who become hospitalized with COVID-19, participation in investigational treatment studies is permitted.
6. Has previously received a documented complete two dose series of the BBIBP-CorV vaccine with the second dose having been given at least 180 days prior to study vaccination OR has previously received a documented complete two dose series of the BBIBP-CorV vaccine and a third dose booster of BBIBP-CorV vaccine, with the third dose having been given at least 90 days prior to study vaccination.

Exclusion Criteria:

1. Participation in research involving receipt of investigational products (drug/biologic/device) within 90 days prior to first study vaccination.
2. Has previously received a primary series vaccination or booster dose of any COVID- 19 vaccine other than BBIBP-CorV.
3. Received influenza vaccination within 14 days prior to first study vaccination, or any other vaccine (including COVID-19) within 30 days prior to first study vaccination.
4. Any known allergies to products contained in the investigational product
5. Any history of anaphylaxis to any prior vaccine.
6. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) requiring ongoing immunomodulatory therapy. NOTE: Stable endocrine disorders (eg, thyroiditis, pancreatitis), including stable diabetes mellitus with no history of diabetic ketoacidosis are NOT excluded.
7. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to first study vaccination. NOTE: An immunosuppressant dose of glucocorticoid is defined as a systemic dose

   ≥ 10 mg of prednisone per day or equivalent. The use of topical or intranasal glucocorticoids is permitted. Topical tacrolimus and ocular cyclosporin are permitted.

   Use of inhaled glucocorticoids is prohibited.
8. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to first study vaccination.
9. Active cancer (malignancy) on therapy within 3 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
10. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study.
11. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to the first study vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.
12. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
13. Study team member or immediate family member of any study team member (inclusive of Sponsor, CRO, and study site personnel involved in the conduct or planning of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Utilizing ratio of IgG GMTs and difference in seroconversion rates to compare IgG antibody responses between the vaccines. | On Day 14.
  Comparative IgG antibody responses on Day 14, summarized in terms of the ratio of IgG GMTs and difference in seroconversion rates (SCR; defined as ≥ 4-fold increase from baseline booster dose) between the vaccines. Non-inferiority will be demonstrated if:
  * The lower bound of the two-sided 95% CI on the ratio of the GMTS (GMTNVX-CoV2373/GMTBBIBP-CorV) is ≥ 0.6667, AND
  * The lower bound of the two-sided 95% CI on the difference between the SCRs (SCRNVX-CoV2373 - SCR BBIBP-CorV) is ≥ 10%.
Utilizing Case Report Forms and safety follow up via telephone to measure and assess incidence, duration, and severity of solicited local and systemic adverse events (AEs) | For 7 days following each vaccination.
  All safety analyses will be summarized descriptively by vaccine group using the Safety Analysis Set. To compare the overall safety, the two-sided 95% CIs for the difference of incidence of solicited AEs for 7 days following each vaccination. Recording of solicited and unsolicited AEs may be conducted by electronic data capture (EDC)/reporting. All AEs will be followed until resolution or until clinically stable.
Utilizing Case Report Forms to measure and assess Incidence, duration, severity, and relationship of unsolicited AEs | Through 28 days after the last vaccination.
  All safety analyses will be summarized descriptively by vaccine group using the Safety Analysis Set. 1085BUnsolicited AEs will be coded by preferred term and system organ class using MedDRA and summarized by vaccine group as well as by severity and relationship to booster vaccine. Unsolicited AEs through 28 days after the booster vaccination. Recording of solicited and unsolicited AEs may be conducted by electronic data capture (EDC)/reporting. All AEs will be followed until resolution or until clinically stable.
Utilizing Case Report Forms to measure incidence and relationship of medically attended adverse events (MAAEs), adverse events of special interest (AESIs) (predefined list), and serious adverse events (SAEs) throughout the study. | Throughout the study. Note: Beginning on Day 29, only MAAEs related to the vaccine will be recorded.
  To compare the overall safety of a single booster injection of NVX-CoV2373 with Matrix-M adjuvant with a single booster injection of BBIBP-CorV in participants previously vaccinated with a primary two-dose series of the BBIBP-CorV vaccine. Recording of solicited and unsolicited AEs may be conducted by electronic data capture (EDC)/reporting. All AEs will be followed until resolution or until clinically stable.

SECONDARY OUTCOMES:
Utilizing Plaque Reduction Neutralization Tests (PRNT) to compare neutralizing antibody responses | • PRNT GMTs to the SARS-CoV-2 S protein at Days 0, 14, 28, and 180. • GMFRPost/Pre, defined as the ratio of post-vaccination to pre-vaccination (Day 0) PRNT GMTs within the same treatment arm at Days 14, 28, and 180.
  Objective: Utilize Plaque Reduction Neutralization Tests (PRNT) to compare neutralizing antibody responses to the SARS-CoV-2 rS with Matrix M adjuvant vaccine to antibody responses to the BBIBP-CorV vaccine, both administered as single booster doses, in adult participants ≥18 years of age who were previously vaccinated with a primary two-dose series of BBIBP-CorV.

CONTACTS AND LOCATIONS:
Overall Officials: Nawal Al Kaabi, Principal Investigator — Sheikh Khalifa Medical City
Locations (2):
- United Arab Emirates (2):
  - Cleveland Clinic Abu Dhabi, Abu Dhabi
  - Sheikh Khalifa Medical City (SKMC), Abu Dhabi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Formica N, Mallory R, Albert G, Robinson M, Plested JS, Cho I, Robertson A, Dubovsky F, Glenn GM; 2019nCoV-101 Study Group. Different dose regimens of a SARS-CoV-2 recombinant spike protein vaccine (NVX-CoV2373) in younger and older adults: A phase 2 randomized placebo-controlled trial. PLoS Med. 2021 Oct 1;18(10):e1003769. doi: 10.1371/journal.pmed.1003769. eCollection 2021 Oct. PMID 34597298
- [Background] Guebre-Xabier M, Patel N, Tian JH, Zhou B, Maciejewski S, Lam K, Portnoff AD, Massare MJ, Frieman MB, Piedra PA, Ellingsworth L, Glenn G, Smith G. NVX-CoV2373 vaccine protects cynomolgus macaque upper and lower airways against SARS-CoV-2 challenge. Vaccine. 2020 Nov 25;38(50):7892-7896. doi: 10.1016/j.vaccine.2020.10.064. Epub 2020 Oct 23. PMID 33139139
- [Background] Heath PT, Galiza EP, Baxter DN, Boffito M, Browne D, Burns F, Chadwick DR, Clark R, Cosgrove C, Galloway J, Goodman AL, Heer A, Higham A, Iyengar S, Jamal A, Jeanes C, Kalra PA, Kyriakidou C, McAuley DF, Meyrick A, Minassian AM, Minton J, Moore P, Munsoor I, Nicholls H, Osanlou O, Packham J, Pretswell CH, San Francisco Ramos A, Saralaya D, Sheridan RP, Smith R, Soiza RL, Swift PA, Thomson EC, Turner J, Viljoen ME, Albert G, Cho I, Dubovsky F, Glenn G, Rivers J, Robertson A, Smith K, Toback S; 2019nCoV-302 Study Group. Safety and Efficacy of NVX-CoV2373 Covid-19 Vaccine. N Engl J Med. 2021 Sep 23;385(13):1172-1183. doi: 10.1056/NEJMoa2107659. Epub 2021 Jun 30. PMID 34192426
- [Background] Keech C, Albert G, Cho I, Robertson A, Reed P, Neal S, Plested JS, Zhu M, Cloney-Clark S, Zhou H, Smith G, Patel N, Frieman MB, Haupt RE, Logue J, McGrath M, Weston S, Piedra PA, Desai C, Callahan K, Lewis M, Price-Abbott P, Formica N, Shinde V, Fries L, Lickliter JD, Griffin P, Wilkinson B, Glenn GM. Phase 1-2 Trial of a SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine. N Engl J Med. 2020 Dec 10;383(24):2320-2332. doi: 10.1056/NEJMoa2026920. Epub 2020 Sep 2. PMID 32877576
- [Background] Liu YV, Massare MJ, Barnard DL, Kort T, Nathan M, Wang L, Smith G. Chimeric severe acute respiratory syndrome coronavirus (SARS-CoV) S glycoprotein and influenza matrix 1 efficiently form virus-like particles (VLPs) that protect mice against challenge with SARS-CoV. Vaccine. 2011 Sep 2;29(38):6606-13. doi: 10.1016/j.vaccine.2011.06.111. Epub 2011 Jul 14. PMID 21762752
- [Derived] Toback S, Marchese AM, Warren B, Ayman S, Zarkovic S, ElTantawy I, Mallory RM, Rousculp M, Almarzooqi F, Piechowski-Jozwiak B, Bonilla MF, Bakkour AE, Hussein SE, Al Kaabi N. Safety and immunogenicity of the NVX-CoV2373 vaccine as a booster in adults previously vaccinated with the BBIBP-CorV vaccine. Vaccine. 2024 Mar 7;42(7):1777-1784. doi: 10.1016/j.vaccine.2024.02.037. Epub 2024 Feb 15. PMID 38365482
- See also: FDA Guidance for industry: Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials. — https://www.fda.gov/media/73679/download
- See also: Division of AIDS (DAIDS) table for grading the severity of adult and pediatric adverse events. July 2017 — https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf
- See also: Evaluation of a SARS-CoV-2 vaccine NVX-CoV2373 in younger and older adults — https://doi.org/10.1101/2021.02.26.21252482
- See also: NVX-CoV2373 vaccine protects cynomolgus macaque upper and lower airways against SARS-CoV-2 challenge — https://doi.org/10.1101/2020.08.18.256578
- See also: First-in-Human Trial of a SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine. — https://doi.org/10.1101/2020.08.05.20168435
- See also: Chimeric severe acute respiratory syndrome coronavirus (SARS-CoV) S glycoprotein and influenza matrix 1 efficiently form virus-like particles (VLPs) that protect mice against challenge with SARS-CoV. Vaccine — https://doi.org/10.1016/j.vaccine.2011.06.111
- See also: WHO 2021: World Health Organization.WHO coronavirus disease (COVID-19) dashboard. [cited 20 January 2021] — https://covid19.who.int/region/euro/country/gb
- See also: WHO 2020b: World Health Organization. Naming the coronavirus disease (COVID-19) and the virus that causes it. World Health Organization COVID-19 Update Information [cited 28 December 2020]. — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/technical-guidance/naming-the-coronavirus-disease-(covid-2019)-and-the-virus-that-causes-it
- See also: WHO 2020c: World Health Organization. WHO Coronavirus Disease (COVID-19) Dashboard [cited 28 December 2020] — https://covid19.who.int/